CLINICAL TRIAL: NCT02595281
Title: Determination of the Interest of HE4 as a Relapse Biomarker in Ovarian Cancers Stages IIIb, IIIc and IV After Neo-adjuvant Chemotherapy and Surgery.
Brief Title: HE4 as a Relapse Biomarker in Ovarian Cancers
Acronym: PRONOV4IR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01511-46
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian Carcinoma; neoadjuvant; ROMA; Ca125; HE4; biomarker
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study arm (Experimental)
  Interventions: Other: Experimental arm

INTERVENTIONS:
Other: Experimental arm — Serum samples are collected:
  * at each neoadjuvant chemotherapy cycle
  * before surgery
  * at each adjuvant chemotherapy cycle
  * at each injection of bevacizumab as maintenance therapy
  * stop at the progression or after 24 months post chemotherapy

SUMMARY:
HE4 is a more sensitive marker than CA-125 in patients with ovarian cancers. The interest of serum HE4 before surgery has been demonstrated to predict overall survival and its interest has also been shown in combination with CA-125 (ROMA algorithm) to identify high risk patients. To date, no study shows clearly the predictive potential of serum HE4 as an early relapse biomarker in ovarian cancers.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian adenocarcinoma stage IIIa, IIIb or IV pleural, cytologically or histologically proven
* Patient scheduled to undergo neoadjuvant chemotherapy based on platinum followed by surgery and adjuvant chemotherapy
* Age ≥ 18 years .
* Performance status ECOG > or = 2
* Adequate haemoglobin rate ≥ 10 g/dL
* Ability to provide written informed consent
* Patient's legal capacity to consent to study participation

Exclusion Criteria:

* Any previous treatment with platinum for ovarian carcinoma
* Patient with visceral metastases
* Contraindication for blood test
* Contraindication for surgery
* Contraindication for bevacizumab treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the predictive and prognostic value of HE4 marker | 24 months
  Serum concentration of HE4 (pMol) will be analysed at each visit

SECONDARY OUTCOMES:
Compare the evolution of HE4 and CA-125 serum concentration | 24 months
  Serum concentration of HE4 and CA-125 (pMol) will be analysed and compared at the time of diagnosis, at each neoadjuvant chemotherapy cycle, before the surgery, and at each chemotherapy cycle
Evaluate the progression-free survival at 18 months | 24 months
  HE4 and CA125 will be compared with the rate of progression-free survival
Evaluate the quality of surgery | 24 months
  HE4 and CA125 will be compared with completeness of cancer resection score (CCR score).

CONTACTS AND LOCATIONS:
Overall Officials: Céline Gavoille, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (7):
- France (7):
  - BENGRINE-LEVEVRE Leïla, Dijon, Centre Georges François Leclerc
  - DEMARCHI Martin, Strasbourg, Centre Paul Strauss
  - LONGO Raphaelle, Metz, CHU Metz Thionville
  - KURTZ Jean-Emmanuel, Strasbourg, Hôpital Civil
  - KALBACHER Elsa, Besançon, Hôpital Jean Minjoz
  - GAVOILLE Céline, Vandœuvre-lès-Nancy, Institut de Cancérologie de Lorraine
  - SAVOYE Aude-Marie, Reims, Institut Jean Godinot